CLINICAL TRIAL: NCT02808234
Title: A Single-arm, Prospective, Multi-center Study of Nucel® in Patients Receiving Interbody Fusion for One and Two Level Degenerative Disease of the Lumbar Spine
Brief Title: Study of Nucel for One and Two Level Lumbar Interbody Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nucel-2015-03
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spondylosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nucel treatment group (Other): One or two level lumbar interbody fusion surgery with Nucel
  Interventions: Procedure: One or two level lumbar interbody fusion surgery; Other: Nucel

INTERVENTIONS:
Procedure: One or two level lumbar interbody fusion surgery — One or two level lumbar interbody fusion surgery with allograft derived from human amnion and amniotic fluid.
Other: Nucel — Allograft derived from human amnion and amniotic fluid

SUMMARY:
The study is a prospective non-randomized multi-center feasibility clinical trial to establish the safety and efficacy of the Nucel® allograft tissue for use in lumbar interbody fusion procedures.

DETAILED DESCRIPTION:
Two hundred non-randomized subjects will participate in the study at up to ten clinical sites in the United States. Participants will be between 18 and 75 years of age. All subjects will have been established with lumbar spine disease at one or two levels of the lumbar spine that requires lumbar interbody fusion procedure as per the opinion of the treating surgeon. The diseases included in the study are spondylosis, degenerative disc disease and spondylolisthesis. All subjects who meet the inclusion criteria and do not meet the exclusion criteria and who elect to participate and sign the informed consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 75 years of age
2. Have clinical and/or radiological evidence of stenosis, spondylolisthesis, spondylosis or degenerative disc disease, or at either one or two levels of lumbar spine.
3. In the opinion of the treating surgeon, must already be a qualified candidate for interbody lumbar fusion surgery with supplemental fixation.
4. Be likely to return for regular follow-ups until the end of the study period.
5. Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria:

1. Previous lumbar spine fusion surgery at operative level.
2. Back pain due to acute trauma.
3. Clinical, laboratory and/or radiological evidence of back pain secondary to acute or chronic infection, malignancy, other space occupying lesions and metabolic bone demineralization diseases (e.g. osteomalacia, gout, Paget's disease etc.)
4. No chronic steroid or chronic prescription NSAID use within three (3) months prior to surgery.
5. Any active malignancy, infectious process, or documented chronic autoimmune disease.
6. Any other concurrent medical disease or treatment that might impair normal healing process.
7. Recent history (within past 6 months) of any chemical or alcohol dependence.
8. Morbid obesity (BMI > 40).
9. Currently a prisoner.
10. Currently experiencing a major mental illness (psychosis, schizophrenia, major affective disorder) which may indicate that the symptoms are psychological rather than of physical origin.
11. Pregnancy at the time of enrollment or planned pregnancy, which would interfere with follow-up imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fusion rate using non-contrast CT of the lumbar spine | 2 years
  Fusion will be assessed 2 years by independent radiologist using alpha-numeric grading scale to quantify bone growth and supplemental fixation quality

OTHER OUTCOMES:
Neurologic Exam | 2 years
  Physician conducted neurological exam
Visual Analogue Scale | 2 years
  Patient health outcome survey
Oswestry Low Back Pain Disability Index | 2 years
  Patient health outcome survey
SF-12 health survey | 2 years
  Patient health outcome survey

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Nunley, MD, Principal Investigator — Spine Institute of Louisiana
Locations (3):
- United States (3):
  - Florida Orthopaedic Insitute, Tampa, Florida
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Carolina Neurosurgery & Spine, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No